CLINICAL TRIAL: NCT03352583
Title: Effects of Evening Casein Protein Consumption on Body Composition and Performance
Brief Title: Effects of Casein Timing on Body Composition and Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Responsible Party: Principal Investigator, Jordan Joy, Graduate Research Assistant, Texas Woman's University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18896
Record Dates: First submitted 2017-11-16; First posted 2017-11-24 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Body Composition
MeSH Terms: interventions — Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Day (Active Comparator): Group receives casein protein during the day (greater than 6 hours before bed).
  Interventions: Dietary Supplement: Protein
- Night (Experimental): Group receives casein protein immediately before going to bed.
  Interventions: Dietary Supplement: Protein

INTERVENTIONS:
Dietary Supplement: Protein — 40g calcium caseinate

SUMMARY:
This study will investigate the effects of night time versus day time casein supplementation on body composition and athletic performance. Participants will consume the protein supplements daily while participating in a supervised, periodized resistance training program.

DETAILED DESCRIPTION:
In a randomized, double-blind, placebo-, exercise- and diet-controlled design, 60 subjects will participate in a 10-week study to determine the influence of selective protein timing on body composition, metabolic, and performance adaptations to resistance training. Diets will be individually standardized using the Cunningham equation adjusted for activity level to determine total maintenance calories. Carbohydrates, fats, and proteins will represent 50, 25, and 25 percent of the determined total calories. Diet counseling will occur weekly until stabilized and biweekly thereafter to ensure compliance with food and fluid intake. Protein will be distributed throughout the day as >0.30g/kg bw/meal for breakfast, lunch, and dinner. Resistance training sessions will be supervised by research staff and occur 4 times per week and begin between 7 am and 5pm. Exercises will consist of single- and multi-joint exercises for all major muscle groups (legs, chest, back, shoulders, core, and arms), be performed for 3-5 sets of 1-20 repetitions with 1-5 minutes rest between sets, and each muscle group will undergo 72-96 hours rest between training sessions within the periodized program. Protein supplements. In the treatment group, the casein supplement (40g calcium caseinate dissolved in water) will be consumed as the last meal (>2h following previous meal) before bed and the placebo (40g maltodextrin dissolved in water) either before resistance training, if training after 10am, or after resistance training, if before 10am. The control group will alternate consumption times of the casein supplement and placebo. The supplement (treatment group) or placebo (control group) will not be consumed within 3 hours of beginning or ending resistance training, nor will it be consumed within 3 hours of the first meal following waking. All groups will be provided with 0.30g/kg bw whey protein isolate immediately following training to facilitate recovery. Supplements will be consumed at a similar time of day on non-training days.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* trained (exercises 2-5 days per week for previous 1-3 years)
* maintains regular sleep patterns (7-9 hours per night weekly average)

Exclusion Criteria:

* use of ergogenic aids or medicines known to influence outcomes
* data will be excluded if a participant is <80% compliant with diet and training interventions
* consumes greater than or equal to 12 alcoholic beverages per week
* tobacco use
* dairy allergy

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2016-11-18 (Actual); Study Completion 2016-11-18 (Actual)

PRIMARY OUTCOMES:
Changes in lean soft tissue | pre to post over 10 weeks
  estimation of muscle mass by DXA
Changes in squat 1 repetition maximum | pre to post over 10 weeks
  measure of lower body strength
Changes in bench press 1 repetition maximum | pre to post over 10 weeks
  measure of upper body strength

SECONDARY OUTCOMES:
changes in fat mass | pre to post over 10 weeks
  estimation of body fat by DXA
changes in percent body fat | pre to post over 10 weeks
  estimation of body fat by DXA
changes in quadriceps cross-sectional area | pre to post over 10 weeks
  measure of muscle hypertrophy
changes in quadriceps muscle thickness | pre to post over 10 weeks
  measure of muscle size

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Woman's University, Denton, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Joy JM, Vogel RM, Shane Broughton K, Kudla U, Kerr NY, Davison JM, Wildman REC, DiMarco NM. Daytime and nighttime casein supplements similarly increase muscle size and strength in response to resistance training earlier in the day: a preliminary investigation. J Int Soc Sports Nutr. 2018 May 15;15(1):24. doi: 10.1186/s12970-018-0228-9. PMID 29764464